CLINICAL TRIAL: NCT02874144
Title: A Phase 2A, Single-Center, Randomized, Placebo-Controlled, Double-Blind Study to Assess the Efficacy of an Anti-Inflammatory Agent in Patients With Sinusitis
Brief Title: Anti-Inflammatory Agent in Sinusitis
Acronym: E1416
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Anju Peters, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E1416 Sinus
Record Dates: First submitted 2016-07-26; First posted 2016-08-22 (Estimated); Results first posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Nasal Polyps
MeSH Terms: conditions — Nasal Polyps | interventions — MeRho-Az compound; Biomarkers; Mometasone Furoate; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZ Compound (Experimental): 40 mg 12 weeks TID po
  Interventions: Drug: AZ compound; Other: Collection of Biological Specimens; Drug: Intranasal corticosteroid
- Placebo (Placebo Comparator): 40 mg 12 weeks TID po
  Interventions: Other: Collection of Biological Specimens; Drug: Intranasal corticosteroid; Drug: Placebo

INTERVENTIONS:
Drug: AZ compound — 40 mg three times daily po for 12 weeks
  Arms: AZ Compound
Other: Collection of Biological Specimens — collection of biomarkers for analysis of nasal disease
  Other Names: Biomarkers
Drug: Intranasal corticosteroid — QD Nasal Spray
  Other Names: Nasal Steroid (Nasonex, Flonase)
Drug: Placebo — looks like AZ compound, made by same company, double blind. 40 mg three times daily po for 12 weeks
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of an anti-inflammatory agent compared with placebo in relieving signs and symptoms of disease in patients with sinusitis.

DETAILED DESCRIPTION:
This is a Phase 2a, single-center, randomized, placebo-controlled, double-blind study that includes 12 weeks of treatment with experimental drug anti-inflammatory agent or placebo TID administered orally.

All subjects will be ≥18 years, have sinusitis with persistent symptoms despite standard of care treatment, and have failed a course of steroids in the past.

ELIGIBILITY:
Inclusion Criteria:

1. Females must have a negative urine pregnancy test at screening unless documented to have a hysterectomy or be postmenopausal.

Exclusion Criteria:

1. Inability or unwillingness of a participant to give written informed consent or comply with study protocol
2. Use of any investigational drugs within 30 days of screening.
3. Acute infection needing antibiotic treatment at screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anju T Peters, MD, Principal Investigator — Northwestern University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Price CPE, Guo A, Stevens WW, Cousens L, Vu TT, Suh LA, Erickson KA, Conley D, Grammer LC, Kern RC, Tan BK, Kato A, Schleimer RP, Smith SS, Welch KC, Peters AT. Efficacy of an oral CRTH2 antagonist (AZD1981) in the treatment of chronic rhinosinusitis with nasal polyps in adults: A randomized controlled clinical trial. Clin Exp Allergy. 2022 Jul;52(7):859-867. doi: 10.1111/cea.14158. Epub 2022 May 18. PMID 35524339

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AZ Compound | Placebo
Started | 22 | 21
Completed | 19 | 16
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- AZD + INCS: AZD1981 40 mg 3 times a day orally, added to 2 sprays daily of intranasal corticosteroid (INCS) spray for 12 weeks.
- PLACEBO + INCS: Placebo 3 times a day orally added to 2 sprays daily of intranasal corticosteroid (INCS) spray for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | AZD + INCS | PLACEBO + INCS | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (13) | 47 (12) | 46 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 14 | 8 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 16 | 14 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: TOTAL POLYP SCORE (TPS)
Description: Measure Description:
  Measurement of Primary outcome- 0-4 scale in each nostril, total is 8. The total polyp score is the sum of the right and left nasal polyp score. Maximum is 8, minimum is 0. Higher score indicates worse disease. 0 =No polyps 1=Small polyps in the middle meatus not reaching below the inferior border of the middle turbinate 2=Polyps reaching the lower border of the middle turbinate or polyp medial to the middle turbinate 3 = Large polyps reaching the lower border of the inferior turbinate 4 =Large polyps causing complete obstruction.
  The primary outcome measured change in polyp size and secondary outcomes included change in radiographic severity of sinus disease, quality of life, and nasal symptoms as measured by Sino Nasal Outcome Test-22 (SNOT-22) and sense of smell by Brief Smell Identification Test (B-SIT) at 12 weeks in the AZD1981 group vs. the placebo. These were done at the baseline visit and the Week 12 visit.
Time Frame: Baseline and Week 12
Population: The primary outcome was the mean change from baseline to 12 weeks in the size of nasal polyps as measured by the total polyp score in the AZD1981 treated group compared to the placebo-treated group.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- AZD + INCS: AZD1981 40 mg three times a day , added to 2 sprays daily of intranasal corticosteroid (INCS) spray for 12 weeks.
- PLACEBO + INCS: Matched Placebo (1:1 randomization) three times a day added to 2 sprays daily of intranasal corticosteroid (INCS) spray for 12 weeks.
Arm/Group | AZD + INCS | PLACEBO + INCS
Number analyzed (Participants) | 22 | 21
units on a scale | 4.67 (0.38) | 5.24 (0.36)
Statistical Analysis 1: Comparison: AZD + INCS vs PLACEBO + INCS; We used baseline scores to track change to follow-up scores and used a difference-in-differences (D-I-D) statistical approach to compare the change over time compare relative rate of change over time between scores within the treatment group (AZD1981 plus INCS) and within the to scores within the placebo group (INCS treatment only); Test type: Superiority — intention-to-treat with participants analyzed according to a randomly assigned treatment group irrespective of compliance; p < 0.05, Regression, Linear — The reported p-value was calculated, and is not attempting to indicate the threshold for statistical significance; Slope = 0, Standard Error of Mean 0; For inflammatory mediator analyses, data were reported as mean (SEM) with statistical significance determined by Kruskal-Wallis test
Statistical Analysis 2: Comparison: AZD + INCS vs PLACEBO + INCS; The trial design is a continuous outcome superiority trial with primary efficacy outcome measures of change in Total Polyp Score (TPS) comparing AZD to placebo arm from V1 to V5. Total polyp score is a standardized method for assessing nasal polyp size by endoscopy, based on a scale of 1-4 per side. Inclusion criterion for this study is a TPS of ≥4 with a maximum of 8 and a standard deviation ± 2. A clinically meaningful effect is considered to be a decrease in total polyp score of 1.5; Test type: Superiority — This was a superiority trial. We used repeated-measures linear regression using the mixed procedure to calculate means for each outcome by visits and treatment status. We used baseline scores to track change to follow-up scores and used a difference-in-differences (D-I-D) statistical approach to compare the change over time between scores within the treatment group (AZD1981 plus INCS) to scores within the placebo group (INCS treatment only); p < 0.05, repeated-measures linear regression — No, the p-value was not adjusted for multiple comparisons; We used repeated-measures linear regression using the MIXED procedure to calculate means (SEMS) for each outcome by visits and treatment status; Mean Difference (Final Values) = -20 — Our study did not include at relative risk

2. Primary Outcome: Sinus CT Scan Scores by Lund-Mackay Scores
Description: Measurement of secondary outcome: sinus CT scan scores by Lund-Mckay scores. We measured sinus radiographic severity with Lund-Mackay scores of 0 to 24. 0 was the least severe and 24 was the most severe. This secondary outcomes included change in radiographic severity of sinus disease, as measured by sinus CT scan scores at baseline and 12 weeks in the AZD1981 group vs. the placebo group.
Time Frame: Baseline and Week 12
Population: The secondary outcome was the mean change in Lund-Mackay scores of sinus CT scans from baseline to 12 weeks in the AZD1981 treated group compared to the placebo-treated group.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | AZD + INCS | PLACEBO + INCS
Number analyzed (Participants) | 22 | 21
units on a scale
  Visit 1 (Baseline) | 17.44 (1.38) | 15.53 (1.43)
  Visit 5 (12 weeks) | 18.25 (1.1) | 16.33 (1.14)

3. Primary Outcome: BSIT (Brief Smell Identification Test)
Description: Measurement of secondary outcome- BSIT (brief smell identification test) is a 12-item test measuring sense of smell. This is a multiple choice test with one correct answer out of four possible answer choices. This test features distinct types of smells. Minimum score: 0/12, which indicates that none of the correct answers were chosen on the 12-item test. Maximum score: 12/12, which indicates that all of the correct answers were chosen on the 12-item test. The higher the score, the better the outcome. Only one out of the four possible answer choices for each multiple choice question is correct. There are no subscales.
  This secondary outcome measures sense of smell by Brief Smell Identification Test (B-SIT) at baseline (visit 1) and 12 weeks (visit 5) in the AZD1981 group vs. the placebo group.
Time Frame: Baseline and Week 12
Population: The secondary outcome was the mean change from baseline to 12 weeks of BSIT scores in the AZD1981 treated group compared to the placebo-treated group.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | AZD + INCS | PLACEBO + INCS
Number analyzed (Participants) | 22 | 21
units on a scale
  Visit 1 (Baseline) | 5.75 (0.81) | 5.20 (0.88)
  Visit 5 (12 weeks) | 6.92 (1.12) | 5.80 (1.22)

4. Secondary Outcome: SNOT-22 (Sino-Nasal Outcome Test-22) Score
Description: Measurement of secondary outcome- the SNOT-22 test contains 22 items regarding patient-reported outcomes of sino-nasal symptom severity on a 0-5 scale for each item. 0 is no problem and 5 is problem as bad as it can be, so higher values represent a worse outcome than lower values. The subscale is 0 - 5 of each of the 22 items and the total score is the sum of the subscales of all 22 items. The minimum total score is 0/110. The maximum total score is 110/110.
  This secondary outcome measured change in patient-reported outcomes of nasal symptoms as measured by Sino Nasal Outcome Test-22 (SNOT-22) over 12 weeks in the AZD1981 group vs. the placebo group.
Time Frame: Baseline and Week 12
Population: This secondary outcome was the mean change from baseline to 12 weeks in sinonasal symptoms detailed in the SNOT-22 as measured by the total polyp score in the AZD1981 treated group compared to the placebo-treated group.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | AZD + INCS | PLACEBO + INCS
Number analyzed (Participants) | 22 | 21
units on a scale
  Visit 1 (baseline) | 33.73 (5.17) | 40.41 (5.01)
  Visit 5 (12 weeks) | 26.07 (4.94) | 36.13 (4.78)

5. Secondary Outcome: Visual Analog Scale (VAS)
Description: Measurement of secondary outcome- 0 to 10 scale bilaterally that measures how subjective sinus symptom severity, with 0 being the least troublesome to 10 being the most troublesome over 12 weeks in the AZD1981 group vs. the placebo group.
Time Frame: Baseline and Week 12
Population: The secondary outcome was the mean change from baseline (visit 1) to 12 weeks (visit 5) of the VAS scores in the AZD1981 treated group compared to the placebo-treated group.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | AZD + INCS | PLACEBO + INCS
Number analyzed (Participants) | 22 | 21
units on a scale
  Visit 1 | 5.57 (2.59) | 5.70 (2.60)
  Visit 5 | 4.75 (2.66) | 4.74 (2.66)

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed every 2 weeks for the first month, then every 4 weeks for 12 weeks and during a 4 week washout period, an average of 5 months.
Description: AE and SAE information was collected under GCP and specific IRB guidelines. All patients were assessed for adverse effects every 2 weeks for the first month and then every 4 weeks during the 12-week study and during a 4 week washout period by means of adverse events reports, physical examination, and laboratory tests (complete blood counts and renal and hepatic chemistries).
Groups:
- AZ+INCS: AZD1981 40 mg three times a day , added to 2 sprays daily of intranasal corticosteroid (INCS) spray for 12 weeks.
Arm/Group | AZ+INCS | Placebo + INCS
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/22 | 1/21
Other Adverse Events (participants affected / at risk) | 1/22 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZ+INCS (N=22) | Placebo + INCS (N=21)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypersensitivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Blood and lymphatic system disorders
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZ+INCS (N=22) | Placebo + INCS (N=21)
Rash (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — One subject in the AZ group had a hypersensitivity reaction associated with a rash. This stopped with study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/44/NCT02874144/Prot_SAP_000.pdf